CLINICAL TRIAL: NCT02776839
Title: Monocentric Study for Development of a Smartphone Application for Patients With Depressive
Brief Title: Mobile Sensing and Support for Depression
Acronym: MOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Switzerland: ETH (Unknown); Switzerland: Makora (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MOSS
Record Dates: First submitted 2016-05-09; First posted 2016-05-18 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mobile Sensing (Other): This phase of the study is designed to develop the app. due to algorithms the app should lern to detect depressive symptoms
  Interventions: Device: Mobile sensing

INTERVENTIONS:
Device: Mobile sensing
  Other Names: Mobile app

SUMMARY:
The objective of this study is two fold, first to explore the potential of context sensitive intervention delivery to provide in-situ support for people with depressive symptoms, second to explore the detection of daily-life behavior based on smart phone sensor information to identify subjects with a clinically meaningful depression level.

DETAILED DESCRIPTION:
To conduct a very first pilot trial, a monocentric, single-arm clinical study is conducted. The study is approved by the local ethics committee of the Canton of Zurich in Switzerland and the Swiss Agency for Therapeutic Products. It is conducted in full accordance with the Declaration of Helsinki, with all subjects providing their electronic informed consent prior to participation. As the main interest lies in a proof of concept of the proposed MOSS app, emphasis is put on real life conditions. A range of different recruitment channels is used to attract subjects from the general public; they include physical flyers, online posts on relevant online bulletin boards and the Google Play Store.

ELIGIBILITY:
Inclusion Criteria:

* self-declaration of depressive symptoms
* app runs on Android 4.0 and higher
* germen speaking

Exclusion Criteria:

* psychotic symptoms
* bipolar symptoms
* drug or alcohol dependency
* dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - for depression (PHQ-9) | baseline
  subjective depressive symptoms to compare the detected symptoms measured by the app This outcome is needed for the sensing part of the study

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (ZUF-8)- measures client satisfaction with the app | at post (at least 6 weeks after baseline) however some participants will use the app longer than 6 weeks, maximum 6 months
  Client satisfaction with the app is assessed

OTHER OUTCOMES:
Patient Health Questionnaire - for depression (PHQ-9) change | baseline and every other week for at least 6 weeks up to 6 months
  Change of symptoms due to the Support app. As the study is two-fold and also includes a supporting part, this measure is needed for the supporting part of the study

CONTACTS AND LOCATIONS:
Overall Officials: S Weidt, MD, Principal Investigator — University of Zurich